CLINICAL TRIAL: NCT00227864
Title: A Brief Marijuana Intervention for Adolescent Women
Brief Title: A Brief Marijuana Intervention for Adolescent Women - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Stein, MD, PI, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-18954-1; R01DA018954 (NIH); R01-18954-1
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Marijuana Abuse; Sexual Risk Behaviors
Keywords: marijuana; sexual risk
MeSH Terms: conditions — Marijuana Abuse | interventions — Behavior Therapy; Therapeutics

ARMS (2):
- Treatment as Usual (Placebo Comparator): Participants are administered assessments at baseline, 1, 3 and 6 months
  Interventions: Other: Treatment as Usual
- Intervention (Experimental): Participants complete assessments at baseline, 1, 3 and 6 months, and receive a 2-session behavioral intervention at the baseline and 1-month study appointments.
  Interventions: Behavioral: Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy
  Arms: Intervention
Other: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to examine the efficacy of a brief motivational intervention on marijuana use and sex-risk behavior in young women.

DETAILED DESCRIPTION:
This study holds the promise of developing a brief, efficacious intervention to reduce marijuana use and related sexual risk-taking behavior among the large populaton of late adolescent women who are regular marijuana users. In the abscence of intervention, these women are at heightened risk of contracting HIV and other sexually transmitted infections. Therefore it is crucial to develop an intervention that will reduce their marijuana and subsequent sexual risk taking behavior. The intervention employed in this study represents a novel adaptation of interventions that are well-supported with similar populations. If the current intervention is found to be efficacious, it can be readily integrated into a variety of treatment settings, particularly other primary care settings. In addition, this study will contribute valuable information about the relationship between marijuana use and sexual risk taking behavior and about the mechanisms of change in marijuana use in late adolescent women.

Comparison(s): Participants will be assigned, in this 6 month longitudinal study, to an assessment-only group or an assessment plus intervention group. Those in the intervention group will receive 2 motivational intervention sessions during the first 3 months of their study participation.

ELIGIBILITY:
Inclusion Criteria:

current marijuana use; currently sexually active; able to complete the study procedures in English

Exclusion Criteria:

pregnant; alcohol dependence; drug dependence

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 326 (Actual)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Marijuna use | marijuana use at 6 months

SECONDARY OUTCOMES:
Sex-risk behavior | sex-risk behavior at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, M.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Stein MD, Caviness CM, Anderson BJ. Alcohol use potentiates marijuana problem severity in young adult women. Womens Health Issues. 2014 Jan-Feb;24(1):e77-82. doi: 10.1016/j.whi.2013.10.005. PMID 24439950
- [Derived] Caviness CM, Hagerty CE, Anderson BJ, de Dios MA, Hayaki J, Herman D, Stein MD. Self-efficacy and motivation to quit marijuana use among young women. Am J Addict. 2013 Jul-Aug;22(4):373-80. doi: 10.1111/j.1521-0391.2013.12030.x. PMID 23795877
- [Derived] Stein MD, Hagerty CE, Herman DS, Phipps MG, Anderson BJ. A brief marijuana intervention for non-treatment-seeking young adult women. J Subst Abuse Treat. 2011 Mar;40(2):189-98. doi: 10.1016/j.jsat.2010.11.001. Epub 2010 Dec 24. PMID 21185685